CLINICAL TRIAL: NCT05652569
Title: Comprehensive Assessment of Clinical Features and Biomarkers to Identify Patients With Advanced or Metastatic Breast Cancer for Marker Driven Trials in Humans (CATCH)
Brief Title: CATCH: Implementation of Genomics-guided Precision Medicine in Metastatic Breast Cancer
Acronym: CATCH
Status: Recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Other Study IDs: S-164/2017
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Stage IV Breast Cancer; Precision Oncology; Genomics-Guided Biomarker-Stratification; Personalized Oncology; Genomic Profiling
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Profile; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh-frozen biopsy tissue and EDTA-blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Genomic Profiling / Sequencing — Procedure: genomic profiling (Whole-Genome- / Exome-Sequencing + RNA-Sequencing) on metastatic biopsy lesions

SUMMARY:
CATCH is an indication-specific diagnostic platform, which drives the implementation of integrative, genomic profiling for metastatic breast cancer into the clinics. The main objective of this approach is to identify biomarkers and drug targets to guide targeted therapeutic interventions.

Eligible are all metastatic breast cancer patients (independent of gender), irrespective of molecular subtype.

At initial diagnosis of distant metastasis or progress at disease progression, biopsy samples from a prognostic-relevant metastasis are retrieved during standard-of-care procedures for central analyses, together with blood samples. In parallel to all standard-diagnostic measures, genomic and transcriptomic profiling is conducted to infer the underlying biology of the disease and identify patients who might profit from biomarker-guided interventions in clinical trials.

Samples not required for standard-of-care clinical procedures or genomic profiling are systematically collected in a dedicated bio-repository to fuel translational scientific companion programs. The continuously growing comprehensive database serves as an integrative resource for systematic, prospective multidimensional data collection (clinical records, biomaterial, genomic data).

In summary, the overarching goal is to generate a precision oncology platform to i) identify clinically-actionable biomarkers and drug targets that drive genomics-guided therapies and ii) couple the observational, diagnostic registry platform to an increasing number of independent, biomarker-stratified clinical therapy trials (CATCH-GUIDE).

DETAILED DESCRIPTION:
Study Flow

CATCH has the goal to implement personalized oncology workflows into the clinic. The clinical precision oncology core backbone encompasses a streamlined diagnostic end-to-end pipeline:

Patient screening and enrolment: Metastatic breast cancer (mBC) patients at initial diagnosis of locally-advanced-/ distant metastasis and any other clinical progress are screened for eligibility. The treating physician has to obtain written informed consent prior to enrolment.

Collection of biomaterial: Fresh-frozen tumor tissue from progressive prognostic-relevant metastatic lesions is collected during standard-of-care routine procedures at study entry. Consecutive biopsies can be offered at progress. Blood samples are taken at baseline (V1) to account for germline controls and can be sequentially repeated at 3-monthly intervals for monitoring of therapy response.

Processing and analyses of patient samples: Biomaterials are centrally processed (standard histology/IHC and pathology review for tumor content; analyte extraction, QC according to standardized, quality-controlled, accredited workflows (DIN EN ISO/IEC 17025). Analyte extraction on fresh-frozen tissue encompasses DNA, RNA and protein isolation.

Molecular profiling (Sequencing): Genomic profiling (DIN EN ISO/IEC 17025) is centrally processed to ensure standardization and encompasses whole-genome sequencing (WGS) on fresh-frozen tissue biopsies or whole-exome sequencing (WES) on FFPE specimens (in case of unsuccessful biopsy sampling on recent lesion due to low tumor cell content) complemented by RNA-sequencing.

Clinical bioinformatics /Data curation: Tumor- and treatment-relevant genomic aberrations together with standard clinical as well as histopathological parameters are analyzed and put into the clinical context to delineate biomarkers and actionable alterations as well as to tackle the underlying biology of treatment-resistance.

Molecular Tumor Board (MTB): Molecular data and conclusive biomarker profiles are discussed by clinicians, bioinformaticians, molecular biologists, human geneticists and pathologists in a weekly interdisciplinary MTB established at NCT Heidelberg. Treatment-relevant biomarkers and actionable drug targets are validated independently. Therapeutic options are prioritized within a molecular report.

Therapy Implementation: Patients will be informed in detail by the treating physician to discuss potential genetically-tailored treatment options. The major goal is to offer patients further interventional clinical trials and drive assignment towards genomics-guided matched biomarker / drug combinations.

Follow-up / Documentation Schedule: Clinical documentation is conducted by authorized study personal at study entry in a certified electronic case report form (eCRF) and subsequently every 3 months for at least 3 years, at any staging interval or cancer-specific therapy change to generate a comprehensive patient registry. To ascertain comprehensive follow-up, only patients will be enrolled who will be treated locally at the involved trial sites. Molecular data will be systematically collected to drive translational exploratory research projects.

The following data are collected and stored (baseline and follow-up assessments)

* patient identifier /demographics (including sex, age at diagnosis, family history)
* cancer type / medical history / characteristics diagnosis (including date of diagnosis)
* clinical outcome / longitudinal disease assessments: relapse and progression
* genomic and transcriptomic data
* ECOG status
* sample information (e.g. specimen type, tumor histological type, anatomical location, tissue analyses)
* health-related Quality-of-Life (QoL) / Patient-Reported Outcomes (PROs)

Translational scientific companion programs: Excess biomaterial not needed for the diagnostic precision oncology approach can be used for exploratory research (e.g. ex vivo approaches, liquid biopsies, immunophenotyping).

Results / Outcome Evaluation:Molecular data will be analysed and interpreted on complementary levels. Biomarkers and molecular aberrations such as mutations, amplifications and aberrant gene expression are evaluated for their tumor-relevance and clinical potential to assign patients for specific clinical trials with targeted treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Female and male breast cancer patients ≥ 18 or if the legal guardian has agreed to the respective informed consent form (ICF)
* Patients with advanced or metastatic breast cancer (irrespective of clinical parameters such as TNM, subgroups, therapy lines)
* Patients, who agreed to and were able to sign the informed consent form.

Exclusion Criteria:

* Early breast cancer
* Inability to take a tissue bioptic sample due to reasons such as physical location of the lesion or health of the patient
* Any physical or mental handicap or severe comorbidities that would hamper the adequate cooperation with the patient.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advanced-stage / metastatic breast cancer patients (at the time point of progress)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Setup of the molecular profiling diagnostic platform and feasibility of genomic profiling in metastatic breast cancer. | 31/12/2030
  Total number of advanced stage / metastatic breast cancer patients i) eligible for genomic profiling, ii) successfully genomically-profiled tumors, iii) with conclusive biomarker profiles.
Total number of patients eligible for clinical trials and targeted therapies based on clinical characteristics and comprehensive tumor features. | 31/12/2030
  Patients enrolled in subsequent interventional clinical therapy trials.

SECONDARY OUTCOMES:
Secondary outcome measures Building novel therapeutic hypothesis. | 31/12/2030
  To retrieve qualitative and quantitative biomarker-information on the genomic landscape of breast cancer to setup independent biomarker-guided interventional clinical trials (CATCH-GUIDE).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schneeweiss, MD, Principal Investigator — National Center for Tumor Diseases, Heidelberg; Peter Lichter, PhD, Principal Investigator — German Cancer Research Center; Verena Thewes, PhD, Principal Investigator — National Center for Tumor Diseases, Heidelberg
Locations (12):
- Germany (12):
  - University Hospital Augsburg, Augsburg
  - Charité, Berlin
  - University Hospital Köln, Cologne
  - Medical Faculty and University Hospital Carl Gustav Carus, Dresden
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - National Center for Tumor Diseases, Heidelberg
  - Caritas Hospital St. Josef, Regensburg
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No